CLINICAL TRIAL: NCT00614978
Title: Phase 1 Study of the Combination of Lapatinib and Temozolomide for the Treatment of Progressive Brain Disease in HER-2 Positive Breast Cancer
Brief Title: Lapatinib and Temozolomide for the Treatment of Progressive Brain Disease in HER-2 Positive Breast Cancer
Acronym: LAPTEM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: GlaxoSmithKline (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAP111172; EuDRACT 2007-005132-83
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Breast Cancer; Brain Metastases; HER2 Positive
Keywords: HER-2 positive; brain metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Lapatinib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Lapatinib plus temozolomide
  Interventions: Drug: lapatinib and temozolomide

INTERVENTIONS:
Drug: lapatinib and temozolomide — Temozolomide will be given orally for 5 days of every 28 days, at doses of either 100mg/m2/day or 150mg/m2/day or 200mg/m2/day AND Lapatinib will be given orally every day at either 1000mg/day or 1250mg/day or 1500mg/day.
  Other Names: Tykerb

SUMMARY:
Objectives:

Primary - Determine the maximum tolerated dose (MTD) and evaluate the dose limiting toxicities (DLT) of combining lapatinib and temozolomideSecondary - Obtain preliminary information on the clinical anti-tumor activity of lapatinib plus temozolomide on brain metastases secondary to HER-2 positive breast cancer including Objective Response Rate (ORR), Clinical Benefit (CB) and Duration of Response (DR)

Methodology:

Phase I, single-centre, open-label, dose-escalation study of combining lapatinib and temozolomide in HER-2 positive breast cancer patients with progressive brain metastases after surgery or radiotherapy or radiosurgery

Treatment:

Temozolomide will be given orally for 5 days of every 28 days, at doses of either 100mg/m2/day or 150mg/m2/day or 200mg/m2/day AND Lapatinib will be given orally every day at either 1000mg/day or 1250mg/day or 1500mg/day.Sequential cohorts will be escalated in increments according to the dose escalation scheme, and determined by dose limiting toxicities.

DETAILED DESCRIPTION:
Patients selection criteria:

* age 18 - 70 years
* Women with cytologically or histologically proven metastatic breast cancer with recurrent / progressive brain metastases evaluable by MRI, after standard treatment with surgery (at least 3 weeks prior) or WBRT (at least 3 weeks prior) or stereotactic RT (at least 1 week prior); or otherwise deemed as unsuitable for standard treatment in the first instance
* Known HER-2 positive status (immunohistochemistry (IHC) 3+ Fluorescence In Situ Hybridization (FISH) positive )
* Previous chemotherapy (adjuvant and metastatic regimens) allowed
* Previous treatment with trastuzumab allowed (Trastuzumab to be discontinued prior to study entry)
* At least one measurable lesion in the brain, defined as any lesion >5mm in longest dimension on T1-weighted, gadolinium-enhanced MRI
* Expected life-expectancy of more than 3 months
* ECOG performance status of 0, 1 or 2
* Adequate bone marrow, renal and hepatic functionsLVEF
* LVEF 50% measured by echocardiography or MUGA scan
* Concomitant corticosteroids and anti-convulsants for symptomatic brain metastases are allowed

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years
* Women with cytologically or histologically proven metastatic breast cancer with recurrent / progressive brain metastases evaluable by MRI, after standard treatment with surgery (at least 3 weeks prior) or WBRT (at least 3 weeks prior) or stereotactic RT (at least 1 week prior); or otherwise deemed as unsuitable for standard treatment in the first instance
* Known HER-2 positive status (immunohistochemistry (IHC) 3+ Fluorescence In Situ Hybridization (FISH) positive )
* Previous chemotherapy (adjuvant and metastatic regimens) allowed
* Previous treatment with trastuzumab allowed (Trastuzumab to be discontinued prior to study entry)
* At least one measurable lesion in the brain, defined as any lesion >5mm in longest dimension on T1-weighted, gadolinium-enhanced MRI
* Expected life-expectancy of more than 3 months
* ECOG performance status of 0, 1 or 2
* Adequate bone marrow, renal and hepatic functionsLVEF
* LVEF >50% measured by echocardiography or MUGA scan
* Concomitant corticosteroids and anti-convulsants for symptomatic brain metastases are allowed

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Primary - Determine the maximum tolerated dose (MTD) and evaluate the dose limiting toxicities (DLT) of combining lapatinib and temozolomide | 18 months

SECONDARY OUTCOMES:
Obtain preliminary information on the clinical anti-tumor activity of lapatinib plus temozolomide on brain metastases secondary to HER-2 positive breast cancer including Objective Response Rate, Clinical Benefit and Duration of Response | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Evandro de Azambuja, MD, PhD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium